CLINICAL TRIAL: NCT04963114
Title: Art Therapy Program in the Chronic Phase of Stroke: A Feasibility Pilot Study
Brief Title: Art Therapy Program in the Chronic Phase of Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: McGill University (Other); Laval University (Other); Concordia University, Montreal (Other); Université de Montréal (Other)
Responsible Party: Principal Investigator, Marie-Hélène Milot, researcher and principal investigator, Université de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-31-2019-3003 - ART
Record Dates: First submitted 2021-06-16; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Stroke
Keywords: art therapy; perceptual impairment; depression
MeSH Terms: conditions — Stroke; Depression | interventions — Art Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Art therapy (Experimental): art therapy in the form of a one-hour guided tour of art works followed by a two-hour guided creative painting workshop on specific themes such as beauty and wonder and colors and emotions
  Interventions: Behavioral: art therapy

INTERVENTIONS:
Behavioral: art therapy — guided art tour and workshop

SUMMARY:
INTRODUCTION: After stroke, perceptual impairments, such as negative body perception, contribute to social isolation and depression. In the subacute poststroke phase, art therapy is effective in improving depression, self-esteem, and community integration. Yet, no study has explored the effectiveness of art therapy at the chronic stage of a stroke; where motor recovery is slowed, and body image and self-esteem are deeply challenged.

OBJECTIVES: Primary; to assess the feasibility of an art therapy program (ATP) in the chronic phase of stroke. Secondary; to explore the effects of ATP on perceptual impairment (body image/self-esteem), mood and community integration.

METHOD: Nine adults (stroke ≥6 months) will participate in the ATP consisting of a thematic group visit to the Montreal Museum of Fine Arts followed by an art workshop, supervised by an art therapist (7 visits over 4 months). Feasibility will be evaluated by triangulating data from interviews and subject assessment questionnaires and by assessing retention and attendance. The effects of the ATP will be assessed by changes in perceptual and mood impairment questionnaires (Body Image States, Self-Esteem scales, Beck Depression Inventory-Short-Form) and community integration questionnaire (The Community Integration Questionnaire).

EXPECTED RESULTS AND OUTCOMES: The project will confirm the feasibility of ATP to improve perceptual impairment and community integration post-stroke.

ELIGIBILITY:
Inclusion Criteria:

* be in the chronic stroke phase (≥ 6 months since diagnosis)
* present a low score on the self-esteem scale (score < 32/40 on the French-Canadian Self Esteem Scale)
* present mild to moderate degree of depression (score 4 to 15 in the Beck Depression Abbreviated Inventory)

Exclusion Criteria:

* unable to move autonomously and safely on their own
* present aphasia (score < 28/35 in the communication section of the Stroke Impact Scale)
* present severe hemineglect (score > 70% in the Line Cancelation Test)
* present severe spasticity of the hemi-body (score ≥ 3 on the modified Ashworth scale)
* present cognitive impairment (score ≤ 2/5 in the Mini-Cog)

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Retention rate to the art therapy program | within 7 days after completion of the art therapy program
  the number of participants enrolled at the end of the study divided by the number of participants recruited at the beginning of the study
Adherence to the art therapy program | within 7 days after completion of the art therapy program
  the number of art therapy sessions that participants took part in on a total of 7 visits
Participants' acceptability and perceptions of the effects of the art therapy program | within 7 days after completion of the art therapy program
  Individualized semi-structured 50-minute interviews and a 2-hour focus group interview, conducted by a research assistant, gathered information on the participants acceptability of the art therapy program and its effects on their perceptual problems, mood and level of activity

SECONDARY OUTCOMES:
Change in self esteem assessed with the Rosenberg Self-Esteem Scale | baseline and within 7 days after completion of the art therapy program
  The Rosenberg Self-Esteem Scale: The scale comprises 10 items scored on a 4-point Likert scale ranging from strongly agree to strongly disagree. Scoring ranges from zero to 40, with higher scores indicating higher self-esteem
Change in mood assessed with the Beck Depression Abbreviated Inventory | baseline and within 7 days after completion of the art therapy program
  Beck Depression Abbreviated Inventory : The scale comprises 13 items scored on a 4-point continuum scale (0 = least, 3 = most), with a total summed score ranging from 0 to 39. Higher scores correspond to greater depressive severity
Change in body image assessed with the Body Image States Scale | baseline and within 7 days after completion of the art therapy program
  Body Image States Scale: This 6-item questionnaire assesses, among other things, the persons dissatisfaction or satisfaction (from extremely dissatisfied with to extremely satisfied with) their physical appearance, body size, body shape and weight. The measure is the composite mean of the six 9-point items whereas low scores reflect more negative body image states and high scores reflect more positive states
Change in community integration assessed with the Community Integration Questionnaire | baseline and within 7 days after completion of the art therapy program
  Community Integration Questionnaire: It is a 15-item questionnaire that aims to identify participants' level of integration into home, family life, social activity, and productive activity. The overall score, which represents a summation of the scores from individual questions, ranges from 0 to 29 whereas a higher score indicates greater integration, and a lower score reflects less integration.

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No